CLINICAL TRIAL: NCT04908384
Title: Improving Asthma Care Together (IMPACT): A Shared Management Pilot Study for Children With Asthma and Their Parents
Brief Title: Improving Asthma Care Together (IMPACT): A Shared Management Pilot Study
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jennifer Sonney, Assistant Professor, School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010461; KL2TR002317 (NIH); 1R21NR019328 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2021-06-01 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Asthma in Children
Keywords: Self-management; Shared management; mHealth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACT Intervention (Experimental): IMPACT health application and wearable device
  Interventions: Behavioral: Improving Asthma Care Together (IMPACT)
- Usual care control (No Intervention): Usual care control.

INTERVENTIONS:
Behavioral: Improving Asthma Care Together (IMPACT) — IMPACT is a novel health application and wearable device
  Arms: IMPACT Intervention

SUMMARY:
This study aims to iteratively develop, refine and test the Improving Asthma Care Together (IMPACT) Intervention for school-age children (7-11 years) with persistent asthma and their parents.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic conditions of childhood, affecting over six million US children. Asthma treatment relies on self-management including symptom monitoring and response, trigger avoidance, and timely and appropriate medication use. Unfortunately, fewer than 50% of children with asthma are adherent to asthma treatment regimens, leading to increased disease morbidity and mortality and potentially irreversible airway damage.

Children with asthma are missing a voice in their own care. The school-age years (7-11) represent a natural transition in asthma management, as children must assume some responsibility for asthma-related care while they spend increasing time away from parents at school and other extracurricular activities. Yet, existing interventions focus on parents alone and use prescriptive approaches, telling the parent what to "do" to the child to manage their asthma. As a result, current strategies are failing to provide children with asthma and their families the tools they need to manage asthma successfully within the realities of their daily lives.

Using a Human-Centered Design (HCD) framework, the investigators co-designed a tailored asthma shared management mobile health application that pairs the parent and child together as a team and facilitates the intentional transition of some asthma management to the child. The hypothesis is that by involving children in their own care, participants will improve asthma management in the present, but also establish lifelong successful self-management skills. The objective of the proposed study is to pilot test the Improving Asthma Care Together (IMPACT) mobile health application with parent-child dyads. Based on the preliminary data, the central hypothesis is that IMPACT will be effective for delivering a shared asthma management intervention for children and their parents.

ELIGIBILITY:
CHILD Inclusion Criteria:

* Clinician diagnosis of persistent asthma (prescription for daily asthma medication)
* Speak English

PARENT Inclusion Criteria:

* 18 years or older
* Child's primary caregiver
* Able to understand and read English
* Reside with the child 50% or more
* Legal guardian who can consent for child to participate
* Have access to a smart phone and reliable home internet access
* Reported Asthma Responsibility Questionnaire score < or = 2.5 at screening

CHILD Exclusion Criteria:

* Parent report of developmental delay (language < 5 year level)
* Co-morbid cancer, diabetes, attention deficit hyperactivity disorder (ADHD)
* Current asthma exacerbation at the time of recruitment

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer T Sonney, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonney J, Ward T, Thompson HJ, Kientz JA, Segrin C. Improving Asthma Care Together (IMPACT) mobile health intervention for school-age children with asthma and their parents: a pilot randomised controlled trial study protocol. BMJ Open. 2022 Feb 10;12(2):e059791. doi: 10.1136/bmjopen-2021-059791. PMID 35144958

RESULTS

PARTICIPANT FLOW:
Groups:
- IMPACT Intervention Child Participants: IMPACT health application and wearable device - child participants
  Improving Asthma Care Together (IMPACT): IMPACT is a novel health application and wearable device
- IMPACT Intervention - Parent Participants: IMPACT health application and wearable device - parent participants
  Improving Asthma Care Together (IMPACT): IMPACT is a novel health application and wearable device
- Usual Care Control Child Participants: Usual care control - child participants
- Usual Care Control Parent Participants: Usual care control - parent participants
Period: Overall Study
Arm/Group | IMPACT Intervention Child Participants | IMPACT Intervention - Parent Participants | Usual Care Control Child Participants | Usual Care Control Parent Participants
Started | 21 | 21 | 31 | 31
Completed | 17 | 17 | 31 | 31
Not Completed | 4 | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IMPACT Intervention Child Participants: IMPACT health application and wearable device - child participants
- IMPACT Intervention Parent Participants: IMPACT health application and wearable device - parent participants
- Total: Total of all reporting groups
Arm/Group | IMPACT Intervention Child Participants | IMPACT Intervention Parent Participants | Usual Care Control Child Participants | Usual Care Control Parent Participants | Total
Number analyzed (Participants) | 21 | 21 | 31 | 31 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 0 | 31 | 0 | 52
  Between 18 and 65 years | 0 | 21 | 0 | 31 | 52
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 17 | 29 | 76
  Male | 11 | 1 | 14 | 2 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 6 | 6 | 21
  Not Hispanic or Latino | 16 | 17 | 25 | 25 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 2 | 1 | 7 | 6 | 16
  White | 9 | 14 | 15 | 17 | 55
  More than one race | 8 | 1 | 7 | 3 | 19
  Unknown or Not Reported | 1 | 2 | 1 | 2 | 6
Asthma Responsibility Questionnaire [Mean (Standard Deviation); unit: units on a scale] — 10- items, 5-point scale to report asthma management task responsibility. Total score is the mean of all items calculated. Scores range from 1 to 5, with 1= parent takes responsibility all of the time, 3= parent and child share responsibility about equally, and 5 = child takes responsibility all of the time.
  units on a scale | 2.74 (.55) | 2.4 (.61) | 2.69 (.54) | 2.3 (.7) | 2.5 (.51)
Spirometry - FEV1/FVC [Mean (Standard Deviation); unit: percent of predicted] — Spirometry - objective measure of expiratory lung function will be used to evaluate asthma control. Specifically, the forced expiratory volume in one second/forced vital capacity (FEV1/FVC) measure will be used and interpreted according to the national spirometry guideline cutpoints (NAEPP EPR4 report). Scores are presented as a percentage and typically range from 1% to 120% (occasionally higher), with higher scores indicating better asthma control. Note, national asthma guidelines consider >85% to indicate well controlled asthma. Population: Only measured spirometry in child participants.
  percent of predicted
    number analyzed (Participants) | 21 | 0 | 31 | 0 | 52
    (all) | 85.7 (10.5) |  | 78.6 (13.4) |  | 82.9 (12.1)
Childhood asthma control test [Mean (Standard Deviation); unit: units on a scale] — 7 total items--3 parent (5-point scale) and 4 child (3-point scale) to assess asthma control. Parent and child scores are summed, possible range of 7-27, with higher scores indicate better control. One total score reported for child participants. Population: Scale uses a combination of child and parent participants scores for an overall asthma control score. Overall scores reported under child participants.
  units on a scale
    number analyzed (Participants) | 21 | 0 | 31 | 0 | 52
    (all) | 19.8 (3.19) |  | 21.39 (2.65) |  | 20.8 (2.96)
Asthma Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Self-report child (13 items)- or parent/caregiver (13 items)-reported asthma quality of life, scores range from 1-7 per item, a mean of item scores calculated, with higher scores indicating better quality of life.
  units on a scale | 5.67 (.99) | 5.6 (.95) | 5.88 (.57) | 5.8 (.85) | 5.7 (.61)
Medication Adherence [Mean (Standard Deviation); unit: units on a scale] — Medication Adherence Report Scale for Asthma, 10-items, 5-point scale assessing reported child asthma controller medication adherence at baseline. Baseline assessment of medication adherence allows for analyzing change in adherence following the study intervention. Higher adherence suggests better asthma management. Scores are averaged, ranging from 1-5, with higher scores indicating better adherence.
  units on a scale | 3.7 (.78) | 4.1 (.79) | 3.8 (.75) | 4.0 (.62) | 3.9 (.6)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Responsibility Questionnaire Change From Baseline to 8 Weeks
Description: 10- items, 5-point scale to report asthma management task responsibility. Total score is the mean of all items calculated. Scores range from 1 to 5, with 1= parent takes responsibility all of the time, 3= parent and child share responsibility about equally, and 5 = child takes responsibility all of the time.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Child Intervention Group: Child participants assigned to intervention group
- Parent Intervention Group: Parents assigned to intervention group
- Child Control Group: Child participants assigned to control group
- Parent Control Group: Parent participants assigned to control group
Arm/Group | Child Intervention Group | Parent Intervention Group | Child Control Group | Parent Control Group
Number analyzed (Participants) | 21 | 21 | 31 | 31
score on a scale | 2.72 (.14) | 2.72 (.11) | 2.79 (.1) | 2.31 (.08)

2. Primary Outcome: Asthma Responsibility Questionnaire Change From 8 to 16 Weeks
Description: as for outcome 1
Time Frame: 8 and 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Parent Intervention Group: Parent participants assigned to intervention group
Arm/Group | Child Intervention Group | Parent Intervention Group | Child Control Group | Parent Control Group
Number analyzed (Participants) | 17 | 17 | 31 | 31
score on a scale | 2.88 (.13) | 2.63 (.13) | 2.90 (.1) | 2.4 (.1)

3. Primary Outcome: Asthma Management Self-efficacy Change From Baseline to 8 Weeks
Description: 13-items (parent) and 12-items (child), 5-point scale assesses asthma self-efficacy. Scores are averaged with higher scores indicate higher self-efficacy. Possible range of 1-5.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Child - Intervention Group: Child participants assigned to intervention group
- Child - Control Group: Children assigned to control group
- Parent-control Group: Parent participants assigned to control group
Arm/Group | Child - Intervention Group | Parent Intervention Group | Child - Control Group | Parent-control Group
Number analyzed (Participants) | 19 | 19 | 31 | 31
score on a scale | 3.79 (.11) | 4.27 (.09) | 3.74 (.08) | 4.41 (.07)

4. Primary Outcome: Asthma Management Self-efficacy Change From 8 Weeks to 16 Weeks
Description: 13-items (parent) and 12-items (child), 5-point scale assesses asthma self-efficacy. Scores are averaged and higher scores indicate higher self-efficacy. Possible score range of 1-5.
Time Frame: 8 and 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Child - Intervention Group | Parent Intervention Group | Child - Control Group | Parent-control Group
Number analyzed (Participants) | 17 | 17 | 31 | 31
score on a scale | 3.69 (.12) | 4.36 (.1) | 3.49 (.09) | 4.52 (.08)

5. Secondary Outcome: Spirometry - FEV1/FVC Change From Baseline to 8 Weeks
Description: Spirometry - objective measure of expiratory lung function will be used to evaluate asthma control. Specifically, the forced expiratory volume in one second/forced vital capacity (FEV1/FVC) measure will be used and interpreted according to the national spirometry guideline cutpoints (NAEPP EPR4 report). Scores are presented as a percentage and typically range from 1% to 120% (occasionally higher), with higher scores indicating better asthma control. Note, national asthma guidelines consider >85% to indicate well controlled asthma.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: percentage of predicted
Groups:
- IMPACT Intervention - Child: Child participants assigned to intervention group
- Usual Care Control - Child: Child participants assigned to control group
Arm/Group | IMPACT Intervention - Child | Usual Care Control - Child
Number analyzed (Participants) | 19 | 31
percentage of predicted | 85.18 (3.35) | 82.87 (2.39)

6. Secondary Outcome: Spirometry - FEV1/FVC Change From 8 Weeks to 16 Weeks
Description: as for outcome 5
Time Frame: 8 and 16 weeks
Measure: Mean (Standard Error); unit: percentage of predicted
Groups:
- Intervention - Child Participants: Child participants assigned to intervention
- Control - Child Participants: Child participants assigned to control
Arm/Group | Intervention - Child Participants | Control - Child Participants
Number analyzed (Participants) | 17 | 31
percentage of predicted | 85.38 (2.42) | 81.82 (1.73)

7. Secondary Outcome: Childhood Asthma Control Test Change From Baseline to 8 Weeks
Description: 7 total items--3 parent (5-point scale) and 4 child (3-point scale) to assess asthma control. Parent and child scores are summed, possible range of 7-27, with higher scores indicate better control. One total score reported for child participants.
Time Frame: Baseline and 8 weeks
Population: Scale uses a combination of child and parent participants scores for an overall asthma control score. Overall scores reported under child participants.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Control - Child Participants: Child participants assigned to control group
Arm/Group | Intervention - Child Participants | Control - Child Participants
Number analyzed (Participants) | 19 | 31
score on a scale | 12.46 (.37) | 12.78 (.28)

8. Secondary Outcome: Childhood Asthma Control Test Change From 8 Weeks to 16 Weeks
Description: as for outcome 7
Time Frame: 8 and 16 weeks
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- IMPACT Intervention - Child Participants: Child participants assigned to intervention group
Arm/Group | IMPACT Intervention - Child Participants | Control - Child Participants
Number analyzed (Participants) | 17 | 31
score on a scale | 12.93 (.58) | 12.14 (.43)

9. Secondary Outcome: Childhood Asthma Quality of Life Change From Baseline to 8 Weeks
Description: Self-report child (13 items)- asthma quality of life, scores range from 1-7 per item, a mean of item scores calculated, with higher scores indicating better quality of life. Possible score range of 1-7.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | IMPACT Intervention - Child | Usual Care Control - Child
Number analyzed (Participants) | 19 | 31
score on a scale | 5.74 (.15) | 5.97 (.11)

10. Secondary Outcome: Childhood Asthma Quality of Life Change From 8 Weeks to 16 Weeks
Description: as for outcome 9
Time Frame: 8 and 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Child Participants | Control - Child Participants
Number analyzed (Participants) | 17 | 31
score on a scale | 5.56 (.16) | 5.98 (.12)

11. Secondary Outcome: Parent Asthma Quality of Life Change From Baseline to 8 Weeks
Description: Parent/caregiver (13 items)-reported asthma quality of life, scores range from 1-7 per item, a mean of item scores calculated, with higher scores indicating better quality of life. Score range of variable, which required exponential transformation for negatively skewed distribution, was 2.72-43.35, with higher scores indicating worse quality of life.
Time Frame: Baseline and 8 weeks
Population: Means and SEs for this variable reflect an exponential transformation to compensate for a negatively skewed distribution in the raw variable.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- IMPACT Intervention - Parent: Parent participants assigned to intervention
- Control - Parent: Parent participants assigned to control
Arm/Group | IMPACT Intervention - Parent | Control - Parent
Number analyzed (Participants) | 19 | 31
score on a scale | 11.56 (2.7) | 7.08 (1.27)

12. Secondary Outcome: Parent Asthma Quality of Life Change From 8 Weeks to 16 Weeks
Description: Parent/caregiver (13 items)-reported asthma quality of life, scores range from 1-7 per item, a mean of item scores calculated, with higher scores indicating better quality of life. Score range of variable, which required exponential transformation for negatively skewed distribution, was 2.72-345.90, with higher scores indicating worse quality of life.
Time Frame: 8 and 16 weeks
Population: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | IMPACT Intervention - Parent | Control - Parent
Number analyzed (Participants) | 17 | 31
score on a scale | 12.85 (3.29) | 17.44 (10.99)

13. Secondary Outcome: Acceptability of Intervention Measure (Intervention Groups Only)
Description: 4 items (2 for children) using 5-point scale; scores are summed with higher scores indicate higher acceptability. Possible score range of 4-20 for parents, 2-10 for children.
Time Frame: 8 weeks
Population: Child max score of 10; parent max score of 20
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention - Child Participants: Child participants assigned to intervention group
- Intervention - Parent Participants: Parent participants assigned to intervention group
Arm/Group | Intervention - Child Participants | Intervention - Parent Participants
Number analyzed (Participants) | 19 | 19
score on a scale | 8 (1.26) | 14.42 (3.62)

14. Secondary Outcome: Medication Adherence Change From Baseline to 8 Weeks
Description: Medication Adherence Report Scale for Asthma, 10-items, 5-point scale assessing reported child asthma controller medication adherence at baseline and throughout the study. Higher adherence suggests better asthma management. Scores are averaged, ranging from 1-5, with higher scores indicating better adherence.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Child Intervention Group | Parent Intervention Group | Child Control Group | Parent Control Group
Number analyzed (Participants) | 19 | 19 | 31 | 31
score on a scale | 3.20 (.53) | 3.30 (.44) | 3.70 (.39) | 3.25 (.32)

15. Secondary Outcome: Medication Adherence Change From 8 Weeks to 16 Weeks
Description: as for outcome 14
Time Frame: 8 and 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Child Intervention Group | Parent Intervention Group | Child Control Group | Parent Control Group
Number analyzed (Participants) | 17 | 17 | 31 | 31
score on a scale | 3.32 (.65) | 3.04 (.45) | 3.78 (.48) | 3.65 (.33)

16. Secondary Outcome: Feasibility of Intervention (Intervention Group Only)
Description: 4 items (2 for children) using 5-point scale; scores are summed with higher scores indicate higher feasibility. Possible score range of 4-20 for parents, 2-10 for children.
Time Frame: 8 weeks
Population: child score max of 10; parent max score of 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Child Participants | Intervention - Parent Participants
Number analyzed (Participants) | 19 | 19
score on a scale | 8 (1.17) | 14.37 (3.36)

17. Secondary Outcome: System Usability Scale (Intervention Group Only)
Description: System usability scale - 10 items, 5-point scale to determine perceived usability of a system. To calculate the SUS score, first sum the score contributions from each item. Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall value of SU. Total score may range from 0 to 100 with higher scores indicating higher usability. Used only post-intervention.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Child Participants | Intervention - Parent Participants
Number analyzed (Participants) | 19 | 19
score on a scale | 68.95 (14.03) | 62.5 (19.18)

ADVERSE EVENTS:
Time Frame: During entire study period of 12 months
Groups:
- IMPACT Intervention - Child Participants: IMPACT health application and wearable device - child participants
  Improving Asthma Care Together (IMPACT): IMPACT is a novel health application and wearable device
- Usual Care Control - Child Participants: Usual care control group - child participants
- Usual Care Control - Parent Participants: Usual care control group - parent participants
Arm/Group | IMPACT Intervention - Child Participants | IMPACT Intervention - Parent Participants | Usual Care Control - Child Participants | Usual Care Control - Parent Participants
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04908384/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04908384/SAP_001.pdf